CLINICAL TRIAL: NCT06795958
Title: Non-invasive Detection of Acute Cell-mediated Graft Rejection in Pediatric Heart Transplant Recipients: the Role of Cardiovascular Magnetic Resonance
Brief Title: Non-invasive Detection of Acute Cell-mediated Graft Rejection in Pediatric Heart Transplant Recipients
Status: Recruiting | Type: Observational
Sponsor: IRCCS Azienda Ospedaliero-Universitaria di Bologna (Other)
Responsible Party: Sponsor
Other Study IDs: DAGR
Record Dates: First submitted 2024-12-30; First posted 2025-01-28 (Actual); Last update posted 2025-01-28 (Actual); Status verified 2024-12

CONDITIONS: Pediatric Heart Transplant
Keywords: acute cardiac rejection; paediatric heart transplant; endomyocardial biopsy; multiparametric cardiac; magnetic resonance

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Acute cardiac rejection is currently diagnosed by endomyocardial biopsy (EMB), but multiparametric cardiac magnetic resonance (CMR) may be a non-invasive alternative by its capacity for myocardial structure and function characterization. Our primary aim was to determine the utility of multiparametric CMR in identifying acute graft rejection in paediatric heart transplant recipients. The second aim was to compare textural features of parametric maps in cases of rejection versus those without rejection.

DETAILED DESCRIPTION:
Background:

Heart transplantation is the therapy of choice for paediatric end-stage heart failure to improve survival and quality of life. Survival after cardiac transplantation is linked to the occurrence of complications, especially acute rejection. The diagnosis of acute rejection in cardiac transplant recipients requires invasive technique with endomyocardial biopsy (EMB) which has risks and limitations. Cardiovascular magnetic resonance (CMR) is the gold standard imaging modality for assessing cardiac morphology, ventricular volumes, systolic function and myocardial mass. In addition, CMR allows for assessing the activity of inflammatory changes using markers for myocardial oedema, hyperaemia, capillary leak and irreversible injury applying a combination of non-contrast T2 weighted imaging and more recently parametric mapping techniques (T1 and T2 mapping) and gadolinium enhanced technique.

Native T1 values are higher with increased extracellular compartment by fibrosis and oedema. From native and post-contrast T1, it can calculate extracellular volume fraction (ECV) which represents the interstitial volume. Expansion of interstitial volume occurs with diffuse fibrosis, oedema and infiltrative diseases. T1 and T2 mapping sequences accurately diagnoses interstitial oedema and extracellular space expansion and can potentially detect acute allograft rejection. In paediatric heart transplantation, few studies have assessed these mapping techniques. There is a clear need for a non-invasive and accurate method of detecting acute allograft rejection and late graft disfunction in paediatric heart transplant patients. The overall aim of this study was to determine the utility of multiparametric CMR in identifying acute graft rejection in paediatric heart transplant recipients. In secondary analysis, we aimed to compare textural features of parametric maps in cases of rejection versus those without rejection

Population and study design:

This single center, prospective, cross-sectional study includes children and young adults (transplanted when they were ≤ 18 years) who undergo an EMB for routine surveillance. All consecutive and eligible patients without contraindications to contrast-enhanced CMR during the study period are enrolled.

Patient charts are reviewed for data demographics, transplant history (age of the organ donor, time from transplant, ischemia time of the donor heart, immunosuppressive medications) and rejection history (number and severity of all previous episodes of rejection since heart transplant). Hemodynamic measurements from echocardiography (left ventricular -LV- ejection fraction, mitral E/e'), catheterization (right atrial mean pressure, right ventricle -RV- systolic pressure, RV end diastolic pressure -RVEDP-, main pulmonary artery mean pressure, and pulmonary capillary wedge pressure) and CMR (LV and RV end diastolic volume and global longitudinal and circumferential strain) are also included. Hemodynamic measurements listed above are considered markers of graft dysfunction.

RV septal EMB and right catheterization are performed by experienced clinicians via jugular vein. At least four tissue samples are obtained, stained with hematoxylin and eosin and evaluated using light microscopy. Evidence of cellular rejection and antibody mediated rejection on EMB are graded based on the International Society of Heart and Lung Transplantation (ISHLT) guidelines by a hospital pathologist following standard clinical practises. Clinically, rejection is defined based on treatment plan created by transplant team following EMB procedure. At our institution, those cases with Grade 2 o above acute cellular rejection on biopsy receive new rejection treatment including modification to immunosuppressive therapy, intravenous steroids, thymoglobulin, etc. Those cases with Grade 0 or 1 acute cellular rejection on biopsy don't receive any treatment.

Cases are divided into two groups: Group A includes cases with no rejection and no changes made to their treatment regimen (grade 0 and 1); Group B includes cases with Grade 2 o above acute cellular rejection.

Tissue samples are also evaluated for the presence of antibody-mediated rejection (AMR).

CMR is performed using 1,5 Tesla scanner (Philips Ingenia). Images are analysed by an expert radiologist blinded to patient's clinical data and histology results.

A stack of multiphase short axis slices is acquired using the steady state free precession technique for left and right ventricular volumes. Ventricular volumes are extracted from the cine short axis stack in end-diastole and end-systole in the routine clinical fashion using commercially available software (CVI 42). Ventricular volumes are reported as indexed to recipient body surface area. Ejection fraction for both ventricles are calculated using end-diastolic and end-systolic volumes. The presence of late gadolinium enhancement (LGE) is determined qualitatively on standard long-axis (4-chamber, 2-chamber and 3-chamber) and short-axis slices using phase-sensitive inversion-recovery acquisition (PSIR) > 7 min after the administration of 0,1 ml/kg gadobutrol (Gadovist®, Bayer Spa).

A modified Look-Locker inversion recovery sequence (MOLLI) is used to measure native and post-contrast longitudinal relaxation T1 times of myocardium and blood. Images are acquired in diastole at a basal, mid-ventricular and apical level short axis slices orientation before and > 15 min after administration of contrast. Breathholds are used in cooperative patients and all other patients are scanned during free breathing. Longitudinal relaxation times (T1 times) are measured using commercial available software (CVI42 and Portal Philips). Contours are drawn in the interventricular septum, the left ventricular (LV) free wall and in a region encompassing the entire LV myocardium. T1 times in the blood pool are measured in the LV cavity avoiding papillary muscle. The ECV is calculated using pre- and post-gadolinium T1 times of blood and myocardium as well as the patient's hematocrit, obtained immediately before the scan. Myocardial T1-values is determined according to the American Heart Association 17-segment model and drawing ROIs in the septum. A modified GraSE sequence allowing for myocardial T2 mapping in a single breath-hold per slice using ECG-triggered acquisition of a black blood multi-echo series are acquired in diastole at a basal, mid-ventricular and apical level short axis slices orientation.

Transverse relaxation times (T2 times) are measured using commercial available software (CVI42 and Portal Philips) using the same method of contouring and ROIs of T1 mapping.

Statistical analysis Categorical variables are presented as count (percentage) and continous variables as mean ± standard deviation.

CMR data are stratified according to the presence (grade ≥ 2) or absence (grade 0 or 1) of significant acute cellular rejection on EMB.

In order to identify potential differences between cases with and without acute allograft rejection, the two groups are compared using t-student .

Pearson correlation is performed on T1, T2 and ECV values against markers of graft dysfunction, which included hemodynamic data from echocardiography, catheterization and CMR.

A p-value < 0.05 is considered statistically significant. All statistical analyses are performed using SPSS, 25 version (IBM SPSS Statistics 25).

ELIGIBILITY:
Inclusion Criteria:

* children and young adults (transplanted when they were ≤ 18 years) who undergo an EMB for routine surveillance without contraindications to contrast-enhanced CMR

Exclusion Criteria:

* We also don't recruit recipients who were < 3 months post-heart transplantation to reduce the possibility of confounding from ischemia-reperfusion injury that occurs with the heart transplant procedure

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: children and young adults (transplanted when they were ≤ 18 years)
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2023-12-12 (Actual); Primary Completion 2029-06-30 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
To determine the utility of multiparametric CMR in identifying acute graft rejection in paediatric heart transplant recipients | 1 year
  CMR data were stratified according to the presence (grade ≥ 2) or absence (grade 0 or 1) of significant acute cellular rejection on EMB

CONTACTS AND LOCATIONS:
Overall Officials: Valentina Gesuete, MD, Principal Investigator — IRCCS Azienda Ospedaliero-Universitaria di Bologna
Locations (1):
- IRCCS Azienda Ospedaliero-Universitaria di Bologna, Bologna, Italy

IPD SHARING:
Plan to Share IPD: Undecided